CLINICAL TRIAL: NCT00214760
Title: Phase 3 Randomised, Prospective Study Comparing the PMMA and the Resorbable PEGT/PBT Centralizer by the Uncemented BIHAPRO Total Hip Prosthesis
Brief Title: Polymethyl Methacrylate and (PEGT/PBT) Centralizer by the Uncemented BIHAPRO THP
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: On of the liners has been taken from the market
Sponsor: Biomet Nederland BV (Industry)
Collaborators: Atrium Medical Center (Other)
Responsible Party: Meijers, Atrium medisch centrum
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BMBL_2005_01
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2010-02-01 (Estimated); Status verified 2009-11

CONDITIONS: Osteoarthritis
Keywords: Hip prosthesis; Centralizer; Uncemented
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- PGET (Experimental)
  Interventions: Device: PGET
- PMMA (Active Comparator)
  Interventions: Device: PMMA

INTERVENTIONS:
Device: PGET — resolbable liner
  Other Names: resolbable liner
  Arms: PGET
Device: PMMA — cement liner
  Other Names: cement liner
  Arms: PMMA

SUMMARY:
The purpose of this study is to analyse if the alignment of the stem and the number of complications of the new resorbable PEGT/PBT centralizer are comparable to the standard PMMA centralizer during the placement of an uncemented Bihapro hip prosthesis.

DETAILED DESCRIPTION:
For a correct placement and early fixation of an uncemented hip prosthesis, a centralizer is used. Normally, the centralizer is made of PMMA, the same material as bone cement. When a revision is needed, PMMA is difficult to remove, which is one of the reason not to use a cemented hip prosthesis. With a PMMA centralizer, still PMMA will remain in the bone and needs to be removed in case of a revision. PEGT/PBT is a reabsorbable material, which gives stability during the first month after the placement of the hip prosthesis. However, PEGT/PBT is reabsorped afterwards and, therefore, will not interfere with a revision procedure.

The goal of this study is to analyse if the PEGT/PBT is as safe as PMMA in terms of alignment, direct postoperative complications and clinical results.

Therefore, 100 patients indicated for a cementless Bihapro hip prosthesis which have signed an informed consent are included and randomised over the used centralizers using a weighted randomisation method. All patients will be treated equally. The patients are examined preoperatively, 1 day, 6 weeks, 3, 6, 12, 24 en 48 months postoperatively using an X-ray, the Harris hip score and a patient questionnaire, the Womac and SF36.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Diagnosis: Osteoarthritis
* Indicated for a primary hip prosthesis

Exclusion Criteria:

* Previous hip surgery
* No informed consent
* Active infection in hip
* Immature skeleton
* Rheumatoid arthritis, M. Paget

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2005-05; Primary Completion 2008-08 (Actual); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Alignment | 0,3,6,12,24 months
Complications | all time points

SECONDARY OUTCOMES:
Pain | 0,3,6,12,24 months
Function | 0,3,6,12,24 months

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Bloemsaat-Minekus, PhD, Principal Investigator — Biomet Nederland
Locations (1):
- Atrium medical centre, Heerlen, Netherlands

REFERENCES:
- [Result] Hernandez-Vaquero D, Murcia-Mazon A, Paz-Jimenez J, Alegre-Mateo R, Martinez-Garcia J, Pena-Vazquez J. Behavior of the femoral stem in the Bihapro hip prosthesis. Orthopedics. 1999 Nov;22(11):1049-53. doi: 10.3928/0147-7447-19991101-13. PMID 10580823